CLINICAL TRIAL: NCT07196215
Title: Comparison of Post-operative Pain After Different Root Canal Irrigant Activation Methods in Maxillary Incisors With Symptomatic Irreversible Pulpitis
Brief Title: Comparison of Post-operative Pain After Different Root Canal Irrigant Activation Methods
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RANA AHMAD (Other)
Responsible Party: Sponsor-Investigator, RANA AHMAD, Assistant Professor, Shaheed Zulfiqar Ali Bhutto Medical University
Organization: Shaheed Zulfiqar Ali Bhutto Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TUF/IRB/21/25
Record Dates: First submitted 2025-09-18; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Irriversible Pulpitis; Irrigation; Activation, Patient
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Passive ultrasonic activation (Active Comparator): passive ultrasonic irrigant activation will be performed by using a stainless steel ultrasonic Irrisafe file of size 20 (IRRI S 21/25; VDW, Germany) mounted on ultrasonic unit (Woodpecker Ultrasonic Scaler UDS-J). The file will be kept 2 mm short of working length loosely without binding to the canal. 2.5% NaOCl will be activated for 30 seconds by using a power setting of five.
  Interventions: Procedure: passive ultrasonic activation
- Sonic activation (Active Comparator): In group B, root canals will be filled with 2.5% sodium hypochlorite and medium size tip (red, 25/04) of EndoAcivator (YAHOPE A3, China) will be used keeping it 2 mm short of working length. The activation of irrigant will be done in 2-3 mm vertical strokes for 30 seconds in between each instrumentation
  Interventions: Procedure: sonic activation

INTERVENTIONS:
Procedure: passive ultrasonic activation — passive ultrasonic irrigant activation will be performed by using a stainless steel ultrasonic Irrisafe file of size 20 (IRRI S 21/25; VDW, Germany) mounted on ultrasonic unit (Woodpecker Ultrasonic Scaler UDS-J). The file will be kept 2 mm short of working length loosely without binding to the canal. 2.5% NaOCl will be activated for 30 seconds by using a power setting of five
  Arms: Passive ultrasonic activation
Procedure: sonic activation — root canals will be filled with 2.5% sodium hypochlorite and medium size tip (red, 25/04) of EndoAcivator (YAHOPE A3, China) will be used keeping it 2 mm short of working length. The activation of irrigant will be done in 2-3 mm vertical strokes for 30 seconds in between each instrumentation
  Arms: Sonic activation

SUMMARY:
root canal irrigation protocol

DETAILED DESCRIPTION:
To compare mean post-operative pain intensity at different time intervals (24h and 48h) using visual analogue scale (VAS) in maxillary incisors with symptomatic irreversible pulpitis using two different irrigation activation methods (passive ultrasonic activation and sonic activation using EndoActivator).

ELIGIBILITY:
Inclusion Criteria:

* • Patients in good health with no systemic disease (ASA Class I or II)

  * Age range is between 20 to 50 years.
  * Patients diagnosed with symptomatic irreversible pulpitis in maxillary incisor teeth.
  * Patients who can understand VAS.
  * Patients who give verbal consent to participate voluntarily in the study.

Exclusion Criteria:

* • History of systemic disorder.

  * Pregnant / lactating females (As per medical record/verbally)
  * Patients who had taken preoperative drugs as anti-inflammatory analgesic or antibiotics.
  * Patients with swelling or acute peri-apical abscess.
  * Tooth not suitable for restoration.
  * Periodontally compromised teeth.
  * Retreatment cases.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
pain score on visual analogue scale | 48 hours
  After complete root canal irrigation and preparation, canals will be dried and a temporary dressing of Cavit will be placed. Patients will be reappointed for obturation. VAS scale ranging from 0-10 will be given to patient and will be demonstrated on how to record their pain and which will be recorded by the patient after 24 hours and 48 hours by marking on a chart ranging from 0-10 with 0 = no pain, 1-3 = mild pain, 4-6 = moderate pain 7-10 = severe pain. On 5th day of follow-up, obturation will be done using single cone obturation method

IPD SHARING:
Plan to Share IPD: Yes
outcome measures
Supporting Information: Study Protocol, SAP, ICF
Time Frame: start date: august 2027 end date: december 2027
Access Criteria: principal investigator will have access by contacting corresponding author

REFERENCES:
- [Background] Gundogar M, Sezgin GP, Kaplan SS, Ozyurek H, Uslu G, Ozyurek T. Postoperative pain after different irrigation activation techniques: a randomized, clinical trial. Odontology. 2021 Apr;109(2):385-392. doi: 10.1007/s10266-020-00553-5. Epub 2020 Sep 11. PMID 32915346
- [Background] Narla RK, J RK, Pavuluri TC, P KC, Penumaka R, Nagelli RK. Effect of Different Irrigant Activation Techniques on the Penetration of Calcium Hydroxide, an Intracanal Medicament: An In Vitro Study. Cureus. 2023 Nov 13;15(11):e48768. doi: 10.7759/cureus.48768. eCollection 2023 Nov. PMID 38098913
- [Background] 7. Nivedhitha S. Influence of different irrigant activation techniques in post-operative endodontic pain-a review of literature. Int J Dentistry Oral Sci. 2021;8(5):2659-65.
- [Background] 6. Abou Khalaf Y, Hashem A, Kamel W, Badr M. Postoperative pain after different root canal irrigant activation methods; (randomized clinical trial). Future Dent J. 2021;7(1):1-6.
- [Background] 5. Elzainy P, Hussein W, Hashem A, Badr M. Post-operative pain after different root canal irrigant activation methods in patients with acute apical periodontitis (Randomized Clinical Trial). Open Access Maced J Med Sci. 2022;10(D):331-7.
- [Background] Kumar P, Yadav SK, Chugh VK, Sharma R, Pathak K, Duraisamy A. Comparative Assessment of Postoperative Pain After Three Irrigation Techniques in Single-Rooted Teeth With Symptomatic Irreversible Pulpitis and Symptomatic Apical Periodontitis: A Randomized Controlled Trial. Cureus. 2024 Jul 29;16(7):e65618. doi: 10.7759/cureus.65618. eCollection 2024 Jul. PMID 39205753
- [Background] 3. Salim A, Darrag A, Ghoneim W. Post-operative pain after single-visit endodontic treatment using different root canal irrigation activating techniques. Egypt Dent J. 2021;67(4):3719-30.
- [Background] Sathorn C, Parashos P, Messer H. The prevalence of postoperative pain and flare-up in single- and multiple-visit endodontic treatment: a systematic review. Int Endod J. 2008 Feb;41(2):91-9. doi: 10.1111/j.1365-2591.2007.01316.x. Epub 2007 Oct 23. PMID 17956561
- [Background] Parirokh M, Jalali S, Haghdoost AA, Abbott PV. Comparison of the effect of various irrigants on apically extruded debris after root canal preparation. J Endod. 2012 Feb;38(2):196-9. doi: 10.1016/j.joen.2011.10.027. Epub 2011 Dec 6. PMID 22244635